CLINICAL TRIAL: NCT01736475
Title: A Phase 2/3, Multi-Center, Open Label Study of Efficacy, Safety, and Pharmacokinetics of PEGylated Recombinant Factor VIII (BAX 855) Administered for Prophylaxis and Treatment of Bleeding in Previously Treated Patients With Severe Hemophilia A
Brief Title: Study Investigating a PEGylated Recombinant Factor VIII (BAX 855) for Hemophilia A (PROLONG-ATE Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 261201; 2012-003599-38 (EudraCT Number)
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis (Experimental)
  Interventions: Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method; Biological: PEGylated Recombinant Factor VIII
- On-demand (Experimental)
  Interventions: Biological: PEGylated Recombinant Factor VIII

INTERVENTIONS:
Biological: Antihemophilic Factor (Recombinant) - Plasma/Albumin Free Method — Pharmacokinetic (PK) evaluation of ADVATE
  Other Names: ADVATE
  Arms: Prophylaxis
Biological: PEGylated Recombinant Factor VIII — Pharmacokinetic (PK) evaluation of BAX 855
  Other Names: BAX 855
  Arms: Prophylaxis
Biological: PEGylated Recombinant Factor VIII — Prophylaxis treatment
  Other Names: BAX 855
  Arms: Prophylaxis
Biological: PEGylated Recombinant Factor VIII — On-demand treatment
  Other Names: BAX 855
  Arms: On-demand

SUMMARY:
To assess efficacy and safety, including immunogenicity of BAX 855 administered as prophylaxis and as on-demand therapy in adult and adolescent (12-65 years) previously treated patients (PTPs) with severe hemophilia A To determine the pharmacokinetic (PK) parameters of BAX 855.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant and/or legal representative has/have voluntarily provided signed informed consent
* Participant is 12 to 65 years old at the time of screening
* Participant is male with severe hemophilia A (Factor VIII (FVIII) clotting activity < 1%) as confirmed by central laboratory at screening after the appropriate washout period or a documented FVIII clotting activity <1%
* Participant has been previously treated with plasma-derived FVIII concentrates or recombinant FVIII for ≥150 documented exposure days (EDs)
* Participant is currently receiving prophylaxis or on-demand therapy with FVIII
* Participant is willing and able to comply with the requirements of the protocol

Main Exclusion Criteria:

* Participant has detectable FVIII inhibitory antibodies (≥ 0.6 Bethesda Units (BU) using the Nijmegen modification of the Bethesda assay) as confirmed by central laboratory at screening
* Participant has history of FVIII inhibitory antibodies (≥ 0.4 BU using the Nijmegen modification of the Bethesda assay or ≥ 0.6 BU using the Bethesda assay) at any time prior to screening
* Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease).

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2014-07-17 (Actual); Study Completion 2014-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (72):
- United States (17):
  - University of Colorado, Aurora, Colorado
  - University of Florida, College of Medicine, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Tulane University Medical School, New Orleans, Louisiana
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Palmetto Health, Columbia, South Carolina
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Puget Sound Blood Group, Seattle, Washington
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Clayton, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Hollywood Specialist Centre, Nedlands, Western Australia
- Austria (2):
  - Landes-Frauen-und Kinderklinik Linz, Linz
  - AKH - Medizinische Universität Wien, Vienna
- SHAT of Oncohaematology Diseases, Sofia, Bulgaria
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
- Germany (4):
  - Gerinnungszentrum Rhein-Ruhr, Duisburg, North Rhine-Westphalia
  - Vivantes Klinikum im Friedrichshain - Landsberger Allee, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Werlhof-Institut MVZ, Hanover
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Chaim Sheba Medical Center, Tel Aviv
- Japan (8):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - University of Occupational and Environmental Health Hospital, Kitakyushu-shi, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo-To
  - Ogikubo Hospital, Suginami-ku, Tokyo-To
- Lithuania (2):
  - Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius
  - Children's Hospital, Affiliate of Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Malaysia (3):
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - Pusat Darah Negara, Kuala Lumpur
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewodzki Szpital Specjalistyczny im.M.Kopernika w Lodzi, Lodz
- Sanador SRL, Bucharest, Romania
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Pusan National University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Kyung hee University Hospital at Gangdong, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (4):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska Universitetssjukhuset, Solna, Stockholm
- Universitatsspital Zurich, Zurich, Switzerland
- Tri-Service General Hospital, Taipei, Taiwan
- Ukraine (2):
  - SI V.K.Gusak Emergency and Reconstructive Surgery Institute of NAMSU Center of IT, Donetsk
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Royal Free Hospital, London, Greater London
  - St Thomas' Hospital, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Churchill Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Konkle BA, Stasyshyn O, Chowdary P, Bevan DH, Mant T, Shima M, Engl W, Dyck-Jones J, Fuerlinger M, Patrone L, Ewenstein B, Abbuehl B. Pegylated, full-length, recombinant factor VIII for prophylactic and on-demand treatment of severe hemophilia A. Blood. 2015 Aug 27;126(9):1078-85. doi: 10.1182/blood-2015-03-630897. Epub 2015 Jul 8. PMID 26157075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled (signed informed consent) at 72 sites.
Pre-assignment Details: A total of 159 participants provided informed consent and were screened for study participation, of which there were 21 screen failures. 138 participants were assigned to the prophylactic arm or the on-demand treatment regimen.
Groups:
- Prophylaxis: Twice weekly at a dose of 45 ± 5 IU/kg
- On-demand: 10 to 60 ± 5 IU/kg
Period: Overall Study
Arm/Group | Prophylaxis | On-demand
Started | 121 | 17
Completed | 109 | 17
Not Completed | 12 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Other - Screen failure | 1 | 0
Not completed — Other - Surgical procedure | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Study Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis | On-demand | Total
Number analyzed (Participants) | 121 | 17 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (12.53) | 31.5 (11.05) | 30.0 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 121 | 17 | 138

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR)
Description: Comparisons between prophylactic and on-demand treatment were based on ABR estimates from a negative binomial regression model, taking into account the treatment regimen, target joints and age at screening, and duration of the observation period for efficacy.
Time Frame: 9 months
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Bleeds per year
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 120 | 17
Bleeds per year | 4.3 [3.4 to 5.5] | 43.4 [25.2 to 74.8]
Statistical Analysis 1: Comparison: Prophylaxis vs On-demand; Ratio Annualized Bleeding Rate (ABR) Prophylaxis/On-demand: Prophylaxis treatment w ill be considered to be successful if the upper limit of the 95% CI for the ratio between treatment regimen does not exceed 0.5 (corresponding to a 50% reduction of the mean ABR compared to the on-demand treatment). H01: μ1 ≥0.5*μ2 Ha1: μ1<0.5*μ2 w here μ1 and μ2 are the mean ABRs in on prophylaxis and on-demand, respectively; Test type: Superiority or Other; p < 0.0001, Regression, Negative binomial; Ratio of means = 0.10, 95% CI 2-sided [0.06 to 0.19]

2. Secondary Outcome: Rate of Success of BAX 855 for Treatment of Bleeding Episodes
Description: Success in the control of bleeding was defined as a rating of excellent or good using the Efficacy Rating Scale for Treatment of Bleeding Episodes measured 24 hours after initiation of treatment for the bleeding episode. EXCELLENT: Full relief of pain and cessation of objective signs of bleeding (eg, swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) after a single infusion. No additional infusion is required for the control of bleeding. Administration of further infusions to maintain hemostasis would not affect this scoring. GOOD: Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. FAIR: Probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion. Required more than 1 infusion for complete resolution. NONE: No improvement or condition worsens.
Time Frame: At least 50 exposure days or 6 months (±2 weeks), whichever occurs last, for the prophylaxis arm and 6 months (± 2 weeks) for the on-demand arm.
Population: Full Analysis Set - All bleeding episodes treated with BAX 855 in participants on on-demand and prophylaxis treatment regimens were analyzed as a single group.
Measure: Number (95% Confidence Interval); unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- Participants With a Bleeding Episode: All bleeding episodes treated with BAX 855 in participants on on-demand and prophylaxis treatment regimens.
Arm/Group | Participants With a Bleeding Episode
Number analyzed (Participants) | 81
Number analyzed (Bleeding episodes) | 591
Bleeding episodes | 0.96 [0.91 to 0.98]

3. Secondary Outcome: Average Number of BAX 855 Infusions Needed for the Treatment of Bleeding Episodes
Time Frame: From first exposure to BAX 855 until the end of the study, [at least 50 exposure days or 6 months (±2 weeks), whichever occurs last, for the prophylaxis arm; and 6 months (± 2 weeks) for the on-demand arm].
Population: Participants from the Full Analysis Set who experienced at least one bleeding episode.
Measure: Mean (Standard Deviation); unit: Infusions
Groups:
- Prophylaxis: Break-through bleeds during prophylaxis
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 65 | 17
Infusions | 1.37 (0.80) | 1.21 (0.35)

4. Secondary Outcome: Number of Participants With ≤1, 2, 3, 4, 5, 6, or >6 Month Time Intervals Between Bleeding Episodes or no Bleeding Episodes
Description: Interval between Bleeds in months was calculated as: Observation period for efficacy (in days)/(number of bleeds)*(12/365.2425)
Time Frame: as for outcome 3
Population: Study participants from the Full Analysis Set (FAS) who received BAX855 during the study period. Note: one participant was assigned to the prophylactic arm (thus was included in the FAS) and received only ADVATE during the screening period.
Measure: Number; unit: Participants
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 120 | 17
Participants
  No bleed | 45 | 0
  >6 Months | 5 | 0
  6 Months | 20 | 0
  5 Months | 3 | 0
  4 Months | 0 | 0
  3 Months | 11 | 0
  2 Months | 16 | 0
  ≤1 Month | 20 | 17

5. Secondary Outcome: Weight-adjusted Consumption of BAX 855 - Per Prophylactic Infusion and Pharmacokinetic (PK) Infusion
Time Frame: Prophylactic Infusion: ≥50 exposure days or 6 months (±2 weeks), whichever occurs last. PK Infusion: PK #1 Pre-infusion within 30 minutes; Post-infusion 10 min, and 0.5, 1, 3, 6, 24, 32, 48, 56 hours (h). PK #2 also at Post-infusion 96h
Population: Full Analysis Set (FAS) - Note: data analyzed by subsets of FAS (1) participants who received BAX855 prophylactic infusion or (2) BAX855 pharmacokinetic (PK) participants. - Subset of participants who received BAX855 prophylactic infusion: N= 120 - Subset of BAX855 pharmacokinetic (PK) participants: N=26
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Infusions
Arm/Group | All Study Participants
Number analyzed (Participants) | 137
Number analyzed (Infusions) | 5941
IU/kg
  Per Prophylactic Infusion (N= 5941 Infusions) | 44.51 (4.556)
  Per PK Infusion (N= 50 Infusions) | 45.48 (2.592)

6. Secondary Outcome: Weight-adjusted Consumption of BAX 855 - Per Treatment of Bleeding Episode (BE) and Per BE for Maintenance of Hemostasis
Description: Infusions per bleeding episode for maintenance of hemostasis only includes infusions following the resolution of a bleed to maintain hemostasis.
Time Frame: Treatment of Bleeding Episode (BE): Minor/Moderate BE every 12 to 24 hours until bleeding is resolved; Major BE every 8 to 12 hours until bleeding is resolved. Per BE for Maintenance of Hemostasis: within 48 hours after bleeding episode resolution.
Population: Full Analysis Set (FAS) - Note: data analyzed by subsets of FAS (1) participants who received BAX855 for treatment of BEs (2) BAX855 for Maintenance of Hemostasis. - Subset of participants who received BAX855 for treatment of BEs: N= 92 - Subset BAX855 for Maintenance of Hemostasis participants: N=16
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Bleeds
Groups:
- All Study Participants: All Study Participants who received at least one infusion of BAX855.
Arm/Group | All Study Participants
Number analyzed (Participants) | 137
Number analyzed (Bleeds) | 592
IU/kg
  Per Treatment of BE (N= 592 bleeds) | 37.44 (28.105)
  Per BE for Maintenance of Hemostasis (N=34 bleeds) | 39.29 (34.206)

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: as for outcome 3
Population: Safety Analysis Set (SAS) - All participants treated with BAX 855 were analyzed as a single group (ie on-demand and prophylaxis treatment regimens were analyzed as a single group).
Measure: Number; unit: percent of participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 137
percent of participants
  SAE, Moderate, Unrelated | 0.7
  SAE, Severe, Unrelated | 2.9
  nSAE, Mild, Unrelated | 40.1
  nSAE, Mild, Related | 3.6
  nSAE, Moderate, Unrelated | 19.0
  nSAE, Moderate, Related | 1.5
  nSAE, Unknown Severity, Unrelated | 0.7
  nSAE, Severe, Unrelated | 1.5

8. Secondary Outcome: Immunogenicity - Number of Participants With Positive Inhibitory Antibodies to FVIII, Binding Antibodies to FVIII, PEG-VIII, PEG and Anti-CHO Antibodies at Study Completion/Termination
Description: Number of participants who received BAX855, with immunogenicity data from study completion/termination visit. FVIII = factor VIII; PEG-VIII = polyethylene glycol-factor VIII; Anti-CHO = Anti-Chinese hamster ovary
Time Frame: as for outcome 3
Population: Safety Analysis Set (SAS) - who received BAX855 during the study period. Note: one participant was assigned to the prophylactic arm but did not receive BAX855 (only received ADVATE, during the screening period).
Measure: Number; unit: Participants
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 120 | 17
Participants
  Inhibitory Antibodies to FVIII (N= 112, 14) | 0 | 0
  IgG: Binding Antibodies FVIII (N= 117, 15) | 0 | 0
  IgM: Binding Antibodies FVIII (N= 117, 15) | 0 | 0
  IgG: Binding Antibodies PEG (N= 117, 15) | 0 | 0
  IgM: Binding Antibodies PEG (N= 117, 15) | 0 | 0
  IgG: Binding Antibodies PEG-FVIII (N= 117, 15) | 0 | 1
  IgM: Binding Antibodies PEG-FVIII (N= 117, 15) | 0 | 0
  CHO-Protein Antibodies (N= 117, 15) | 0 | 0

9. Secondary Outcome: Patient Reported Outcomes: Haemo-SYM Questionnaire, Change in Score From Baseline to End of Study
Description: The HAEMO-SYM has two subscales: pain and bleeds. HAEMO-SYM subscale scores are calculated by taking the mean of the items in each subscale and transforming them to a 0 (none or absent) to 100 (very severe) scale. Given that higher scores indicate more severe symptoms on the Haemo-SYM and that the change scores were calculated as the value at study completion minus the value at baseline, a negative change score indicates an improvement (reduction in symptoms). Conversely, a positive change score indicates worsening symptoms.
Time Frame: Baseline; and end of study visit [at least 50 exposure days or 6 months (±2 weeks), whichever occurs last, for the prophylaxis arm and 6 months (± 2 weeks) for the on-demand arm].
Population: Full Analysis Set - Subset of participants with both baseline and study completion HAEMO-SYM scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prophylaxis; On-demand: Participants with both baseline and study completion HAEMO-SYM scores
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 82 | 11
Score on a scale
  Bleed Severity Total Score | -4.17 (17.05) | -4.24 (15.71)
  Pain Severity Total Score | -1.22 (12.50) | -0.17 (11.88)

10. Secondary Outcome: Patient Reported Outcomes - Short Form (SF)-36, Change From Baseline to End of Study
Description: Change from Baseline to End of Study for SF-36 Questionnaire is provided. Scores for individual SF-36 categories range from 0 to 100 with higher scores representing better health. Given that higher scores indicate better health-related quality of life (HRQoL) and that the change scores were calculated as the value at study completion minus the value at baseline, a negative change score indicates a worsening of HRQoL.
Time Frame: as for outcome 9
Population: Full Analysis Set - Subset of participants with both baseline and study completion SF-36 scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prophylaxis; On-demand: Participants with both baseline and study completion SF-36 Scores
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 97 | 12
Score on a scale
  Physical Functioning (N= 97, 12) | 0.49 (5.27) | -2.46 (4.29)
  Role-physical (N= 97, 12) | 1.31 (7.36) | -3.67 (9.01)
  Bodily Pain (N= 97, 12) | 2.08 (8.19) | 0.60 (4.44)
  General Health (N= 96, 12) | 0.40 (6.43) | -0.28 (9.04)
  Vitality (N= 96, 12) | -0.38 (7.43) | 0.26 (9.36)
  Social Functioning (N= 97, 12) | 0.90 (7.54) | -3.18 (6.35)
  Role Emotional (N= 97, 12) | -0.20 (8.46) | 0.65 (7.92)
  Mental Health (N= 96, 12) | 0.09 (7.26) | -3.29 (7.95)
  Physical Component Score (N= 96, 12) | 1.36 (5.76) | -1.58 (4.97)
  Mental Component Score (N= 96, 12) | -0.37 (7.38) | -1.14 (5.03)

11. Secondary Outcome: Pharmacokinetics (Pk) - Plasma Half-life (One-stage Clotting Assay)
Description: Terminal half-life calculated as log_e2/λz where λz is the terminal elimination rate constant. Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: Within 30 minutes prior to start of infusion; and post-infusion at 10, 30 minutes, and 1, 3, 6, 9, 24, 32, 48, 56, 72 (PK2 and PK3 only), and 96 hours (PK2 and PK3 only).
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
hours
  PK-1: ADVATE | 10.40 (2.244)
  PK-2: BAX 855 | 14.30 (3.838)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 16.02 (4.922)

12. Secondary Outcome: Pharmacokinetics (Pk) - Mean Residence Time (One-stage Clotting Assay)
Description: The mean residence time (MRT) w as calculated as total area under the moment curve divided by the total area under the curve starting from the begin of infusion (or the end of infusion if start time is not available). Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
hours
  PK-1: ADVATE | 12.86 (3.044)
  PK-2: BAX 855 | 19.56 (5.315)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 20.65 (4.821)

13. Secondary Outcome: Pharmacokinetics (Pk) - Total Body Clearance (One-stage Clotting Assay)
Description: Clearance in dL/(kg.h) will be calculated as the dose in IU/kg divided by the total area under the curve starting from the begin of infusion (or the end of infusion if start time is not available). Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: dL/(kg*hours)
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
dL/(kg*hours)
  PK-1: ADVATE | 0.04551 (0.021725)
  PK-2: BAX 855 | 0.02760 (0.020288)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 0.02474 (0.008225)

14. Secondary Outcome: Pharmacokinetics (Pk) - Incremental Recovery Over Time (One-stage Clotting Assay)
Description: Incremental recovery (IR) in (IU/dL)/ (IU/kg) calculated as: IR = (Cmax- (C pre-infusion)) / (Dose/kg), where C =concentration. Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
(IU/dL)/(IU/kg)
  PK-1: ADVATE | 2.372 (0.5357)
  PK-2: BAX 855 | 2.493 (0.6944)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 2.297 (0.6377)

15. Secondary Outcome: Pharmacokinetics (Pk) - Area Under the Concentration Versus Time Curve From 0 to Infinity (AUC0-∞) (One-stage Clotting Assay)
Description: Calculated by WinNonlin NCA (Model 201, calculation method: Linear Trapezoidal Linear/Log Interpolation). Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: (IU*hours)/dL
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
(IU*hours)/dL
  PK-1: ADVATE | 1168.0 (425.40)
  PK-2: BAX 855 | 2073.3 (778.41)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 2008.7 (631.53)

16. Secondary Outcome: Pharmacokinetics (Pk) - Apparent Volume of Distribution at Steady State (Vss) (One-stage Clotting Assay)
Description: The apparent volume of distribution at steady state (Vss) will be calculated as: Vss = Clearance * Mean Residence Time. Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
dL/kg
  PK-1: ADVATE | 0.5487 (0.20213)
  PK-2: BAX 855 | 0.4715 (0.14602)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 0.4970 (0.15756)

17. Secondary Outcome: Pharmacokinetics (Pk) - Maximum Plasma Concentration (Cmax) (One-stage Clotting Assay)
Description: Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
IU/dL
  PK-1: ADVATE | 108.45 (26.250)
  PK-2: BAX 855 | 113.68 (30.259)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 103.34 (29.311)

18. Secondary Outcome: Pharmacokinetics (Pk) -Time to Maximum Concentration in Plasma (Tmax) (One-stage Clotting Assay)
Description: Tmax in hours will be defined as the time to reach Cmax. Participants in the pharmacokinetic full analysis set (PKFAS) analysis set received an initial infusion of ADVATE for pharmacokinetic analysis (PK-1) followed by a washout period and an infusion of BAX 855 for a second pharmacokinetic analysis (PK-2). After at least 50 EDs of BAX 855, participants in the PK subgroup received another infusion of BAX 855 for pharmacokinetic analysis (PK-3).
Time Frame: as for outcome 11
Population: Pharmacokinetic full analysis set (PKFAS)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pharmacokinetic Analysis Participants
Number analyzed (Participants) | 26
hours
  PK-1: ADVATE | 0.296 (0.1662)
  PK-2: BAX 855 | 0.397 (0.2632)
  PK-3: BAX 855, After ≥50 Exposure Days (N=22) | 0.467 (0.6044)

19. Secondary Outcome: Change in Vital Signs From Screening - Temperature
Time Frame: Screening, week 2, week 4, exposure day 10-15, month 3, study completion/termination
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Celsius
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 119 | 17
Celsius
  Week 2 (N= 118, 17) | 0.00 [-0.20 to 0.20] | 0.00 [0.00 to 0.20]
  Week 4 (N= 118, 15) | 0.00 [-0.30 to 0.20] | 0.00 [-0.40 to 0.10]
  Exposure day 10-15 (N= 31, 10) | -0.10 [-0.30 to 0.10] | 0.00 [-0.30 to 0.30]
  Month 3 (N= 112, 17) | 0.00 [-0.20 to 0.20] | 0.00 [-0.10 to 0.10]
  Completion/Termination (N= 116, 15) | 0.00 [-0.20 to 0.20] | 0.00 [-0.10 to 0.30]

20. Secondary Outcome: Change in Vital Signs From Screening - Pulse Rate
Time Frame: Screening, week 2, week 4, exposure day 10-15, month 3, study completion/termination
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 118 | 17
beats per minute
  Week 2 (N= 118, 17) | 3.0 [-3.0 to 9.0] | 2.0 [-3.0 to 5.0]
  Week 4 (N= 117, 15) | 2.0 [-4.0 to 10.0] | 2.0 [-5.0 to 4.0]
  Exposure day 10-15 (N= 31, 10) | 3.0 [-3.0 to 10.0] | 4.0 [0.0 to 5.0]
  Month 3 (N= 112, 17) | 2.0 [-5.5 to 6.5] | 1.0 [-6.0 to 8.0]
  Completion/Termination (N= 116, 15) | 2.0 [-6.0 to 8.5] | 3.0 [-5.0 to 10.0]

21. Secondary Outcome: Change in Vital Signs From Screening - Respiratory Rate
Time Frame: Screening, week 2, week 4, exposure day 10-15, month 3, study completion/termination
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: breaths per minute
Arm/Group | Prophylaxis | On-deamand
Number analyzed (Participants) | 118 | 17
breaths per minute
  Week 2 (N= 117, 17) | 0.0 [-1.0 to 1.0] | 0.0 [-1.0 to 2.0]
  Week 4 (N= 118, 15) | 0.0 [-1.0 to 1.0] | 0.0 [-1.0 to 2.0]
  Exposure day 10-15 (N= 31, 10) | 0.0 [-1.0 to 2.0] | 0.0 [-1.0 to 0.0]
  Month 3 (N= 112, 16) | 0.0 [-2.0 to 2.0] | 0.0 [-2.0 to 1.0]
  Completion/Termination (N= 115, 15) | 0.0 [-2.0 to 1.0] | -1.0 [-2.0 to 2.0]

22. Secondary Outcome: Changes in Vital Signs From Screening - Blood Pressure
Description: Systolic Blood Pressure (SBP) Diastolic Blood Pressure (DBP)
Time Frame: Screening, week 2, week 4, exposure day 10-15, month 3, study completion/termination
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 118 | 17
mmHg
  SBP-Week 2 (N= 118, 17) | 0.0 [-7.0 to 6.0] | -2.0 [-9.0 to 7.0]
  SBP-Week 4 (N= 118, 15) | -0.5 [-9.0 to 7.0] | -1.0 [-5.0 to 0.0]
  SBP-Exposure day 10-15 (N= 31, 10) | 0.0 [-5.0 to 4.0] | 3.5 [0.0 to 6.0]
  SBP-Month 3 (N= 112, 17) | 0.0 [-7.0 to 7.5] | -5.0 [-12.0 to 4.0]
  SBP-Completion/Termination (N= 116, 15) | 0.0 [-10.0 to 7.5] | 0.0 [-8.0 to 4.0]
  DBP-Week 2 (N= 118, 17) | 0.0 [-8.0 to 5.0] | -2.0 [-9.0 to 5.0]
  DBP-Week 4 (N= 118, 15) | -0.5 [-6.0 to 5.0] | -6.0 [-12.0 to 7.0]
  DBP-Exposure day 10-15 (N= 31, 10) | 0.0 [-9.0 to 3.0] | -2.5 [-6.0 to 5.0]
  DBP-Month 3 (N= 112, 17) | 0.0 [-7.0 to 7.5] | -4.0 [-9.0 to 5.0]
  DBP-Completion/Termination (N= 116, 15) | 0.0 [-6.0 to 5.0] | -2.0 [-10.0 to 5.0]

23. Secondary Outcome: Changes in Clinical Chemistry Laboratory Assessments From Screening - Albumin and Protein
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 115 | 17
g/L
  Albumin: Week 2 (N= 112, 17) | -1.0 [-2.5 to 1.0] | -1.0 [-2.0 to 0.0]
  Albumin: Week 4 (N= 112, 14) | -1.0 [-3.0 to 0.5] | -1.0 [-2.0 to 0.0]
  Albumin: Month 3 (N= 106, 17) | -1.0 [-3.0 to 1.0] | -1.0 [-2.0 to 1.0]
  Albumin: Completion/Termination (N= 112, 14) | 0.0 [-2.0 to 2.0] | -1.0 [-2.0 to -1.0]
  Protein: Week 2 (N= 115, 17) | -1.0 [-4.0 to 1.0] | -2.0 [-4.0 to 0.0]
  Protein: Week 4 (N= 114, 14) | -1.0 [-4.0 to 1.0] | -2.0 [-5.0 to -1.0]
  Protein: Month 3 (N= 109, 17) | -1.0 [-3.0 to 2.0] | -1.0 [-3.0 to 2.0]
  Protein: Completion/Termination (N= 114, 15) | -1.0 [-3.0 to 2.0] | -1.0 [-4.0 to 0.0]

24. Secondary Outcome: Changes in Clinical Chemistry Laboratory Assessments From Screening - Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase
Description: Alkaline Phosphatase (Alk Phos); Alanine Aminotransferase (Ala Amino); Aspartate Aminotransferase (Asp Amino)
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: Units per Liter
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 115 | 17
Units per Liter
  Alk Phos: Week 2 (N= 115, 17) | -1.0 [-7.0 to 3.0] | -5.0 [-7.0 to 2.0]
  Alk Phos: Week 4 (N= 114, 14) | -4.0 [-9.0 to 2.0] | -4.5 [-10.0 to 1.0]
  Alk Phos: Month 3 (N= 109, 17) | -2.0 [-9.0 to 4.0] | -5.0 [-11.0 to 4.0]
  Alk Phos: Completion/Termination (N= 114, 15) | 0.0 [-9.0 to 6.0] | -5.0 [-9.0 to 1.0]
  Ala Amino: Week 2 (N= 112, 17) | 1.0 [-4.0 to 4.5] | -2.0 [-6.0 to 5.0]
  Ala Amino: Week 4 (N= 112, 14) | 0.0 [-5.0 to 4.0] | -2.5 [-7.0 to 1.0]
  Ala Amino: Month 3 (N= 106, 17) | 1.0 [-6.0 to 5.0] | 1.0 [-4.0 to 12.0]
  Ala Amino: Completion/Termination (N= 112, 14) | -1.0 [-7.0 to 4.0] | 2.5 [-3.0 to 5.0]
  Asp Amino: Week 2 (N= 110, 17) | 0.5 [-2.0 to 5.0] | -1.0 [-6.0 to 2.0]
  Asp Amino: Week 4 (N= 110, 14) | 0.0 [-4.0 to 3.0] | -3.5 [-7.0 to 0.0]
  Asp Amino: Month 3 (N= 103, 17) | 1.0 [-3.0 to 5.0] | 1.0 [-3.0 to 2.0]
  Asp Amino: Completion/Termination (N= 110, 14) | 1.0 [-5.0 to 3.0] | 3.5 [-3.0 to 6.0]

25. Secondary Outcome: Changes in Clinical Chemistry Laboratory Assessments From Screening - Bicarbonate, Chloride, Glucose, Potassium, Sodium, Blood Urea Nitrogen (BUN)
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 115 | 17
mmol/L
  Bicarbonate: Week 2 (N= 111, 16) | 0.10 [-1.60 to 1.40] | 1.10 [-1.50 to 2.60]
  Bicarbonate: Week 4 (N= 110, 13) | 0.40 [-0.90 to 2.40] | 0.10 [-1.50 to 3.00]
  Bicarbonate: Month 3 (N= 111, 16) | 0.60 [-1.30 to 1.90] | 0.60 [-1.30 to 1.75]
  Bicarbonate: Completion/Termination (N= 117, 13) | 1.20 [-0.60 to 2.60] | 2.20 [1.00 to 3.90]
  Chloride: Week 2 (N= 115, 17) | 0.0 [-1.0 to 2.0] | -2.0 [-3.0 to 1.0]
  Chloride: Week 4 (N= 114, 14) | 1.0 [-1.0 to 2.0] | -1.0 [-2.0 to 0.0]
  Chloride: Month 3 (N= 109, 17) | 0.0 [-1.0 to 2.0] | 1.0 [-1.0 to 2.0]
  Chloride: Completion/Termination (N= 114, 15) | 0.0 [-1.0 to 2.0] | -1.0 [-2.0 to 1.0]
  Glucose: Week 2 (N= 112, 17) | -0.10 [-0.55 to 0.55] | -0.30 [-0.80 to 0.20]
  Glucose: Week 4 (N= 112, 14) | 0.10 [-0.40 to 0.70] | -0.05 [-0.50 to 0.50]
  Glucose: Month 3 (N= 106, 17) | 0.00 [-0.50 to 0.50] | 0.10 [-0.50 to 0.30]
  Glucose: Completion/Termination (N= 115, 14) | 0.00 [-0.50 to 0.60] | -0.10 [-0.50 to 0.60]
  Potassium: Week 2 (N= 115, 17) | 0.00 [-0.20 to 0.30] | 0.10 [-0.20 to 0.10]
  Potassium: Week 4 (N= 114, 14) | 0.05 [-0.20 to 0.30] | 0.10 [-0.10 to 0.20]
  Potassium: Month 3 (N= 109, 17) | 0.00 [-0.30 to 0.30] | 0.10 [-0.10 to 0.40]
  Potassium: Completion/Termination (N= 114, 15) | 0.00 [-0.20 to 0.20] | 0.00 [-0.10 to 0.40]
  Sodium: Week 2 (N= 115, 17) | 0.0 [-1.0 to 1.0] | -1.0 [-2.0 to 1.0]
  Sodium: Week 4 (N= 114, 14) | 0.0 [-1.0 to 1.0] | -1.5 [-3.0 to 0.0]
  Sodium: Month 3 (N= 109, 17) | 0.0 [-2.0 to 1.0] | 0.0 [-2.0 to 2.0]
  Sodium: Completion/Termination (N= 114, 15) | -1.0 [-2.0 to 1.0] | -1.0 [-3.0 to 0.0]
  BUN: Week 2 (N= 115, 17) | 0.00 [-0.60 to 0.70] | -0.20 [-0.40 to 0.70]
  BUN: Week 4 (N= 113, 14) | 0.00 [-0.70 to 0.70] | -0.10 [-0.30 to 0.50]
  BUN: Month 3 (N= 109, 17) | 0.30 [-0.30 to 0.90] | -0.40 [-0.70 to 0.30]
  BUN: Completion/Termination (N= 114, 15) | 0.30 [-0.70 to 1.10] | 0.00 [-1.30 to 1.00]

26. Secondary Outcome: Changes in Clinical Chemistry Laboratory Assessments From Screening - Creatinine, and Bilirubin
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: µmol/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 115 | 17
µmol/L
  Creatinine: Week 2 (N= 115, 17) | 0.0 [-7.0 to 4.0] | 1.0 [-3.0 to 4.0]
  Creatinine: Week 4 (N= 114, 14) | 0.0 [-5.0 to 4.0] | 0.5 [-6.0 to 6.0]
  Creatinine: Month 3 (N= 109, 17) | 0.0 [-6.0 to 2.0] | 3.0 [-3.0 to 6.0]
  Creatinine: Completion/Termination (N= 114, 15) | 0.0 [-4.0 to 5.0] | 6.0 [-4.0 to 9.0]
  Bilirubin: Week 2 (N= 109, 17) | 0.00 [-3.00 to 2.00] | -2.00 [-5.00 to 2.00]
  Bilirubin: Week 4 (N= 109, 14) | 0.00 [-2.00 to 2.00] | -0.50 [-5.00 to 3.00]
  Bilirubin: Month 3 (N= 103, 17) | 0.00 [-3.00 to 2.00] | 1.00 [-3.00 to 2.00]
  Bilirubin: Completion/Termination (N= 109, 14) | 0.00 [-3.00 to 2.00] | -0.50 [-2.00 to 3.00]

27. Secondary Outcome: Changes in Hematology Laboratory Assessments From Screening - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, and Leukocytes
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: giga (10^9) cells per liter (Gi/L)
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 109 | 17
giga (10^9) cells per liter (Gi/L)
  Basophils: Week 2 (N= 108, 17) | 0.000 [-0.015 to 0.010] | 0.000 [-0.010 to 0.020]
  Basophils: Week 4 (N= 109, 14) | 0.000 [-0.010 to 0.010] | 0.005 [-0.020 to 0.020]
  Basophils: Month 3 (N= 103, 16) | 0.000 [-0.020 to 0.020] | 0.000 [-0.010 to 0.010]
  Basophils: Completion/Termination (N= 107, 14) | -0.010 [-0.020 to 0.010] | 0.000 [-0.020 to 0.020]
  Eosinophils: Week 2 (N= 108, 17) | 0.010 [-0.020 to 0.050] | 0.030 [0.000 to 0.060]
  Eosinophils: Week 4 (N= 109, 14) | 0.020 [-0.020 to 0.060] | 0.035 [-0.010 to 0.070]
  Eosinophils: Month 3 (N= 103, 16) | 0.010 [-0.040 to 0.050] | 0.010 [-0.005 to 0.050]
  Eosinophils: Completion/Termination (N= 107, 14) | 0.010 [-0.030 to 0.050] | 0.045 [0.010 to 0.080]
  Lymphocytes: Week 2 (N= 108, 17) | -0.005 [-0.215 to 0.140] | 0.280 [-0.070 to 0.640]
  Lymphocytes: Week 4 (N= 109, 14) | -0.060 [-0.240 to 0.210] | 0.175 [0.030 to 0.350]
  Lymphocytes: Month 3 (N= 103, 16) | 0.030 [-0.200 to 0.260] | 0.130 [-0.120 to 0.500]
  Lymphocytes: Completion/Termination (N= 107, 14) | 0.040 [-0.160 to 0.260] | 0.030 [-0.070 to 0.460]
  Monocytes: Week 2 (N= 108, 17) | 0.005 [-0.050 to 0.070] | 0.060 [-0.050 to 0.130]
  Monocytes: Week 4 (N= 109, 14) | 0.020 [-0.060 to 0.050] | -0.010 [-0.070 to 0.040]
  Monocytes: Month 3 (N= 103, 16) | 0.000 [-0.060 to 0.050] | 0.020 [-0.015 to 0.085]
  Monocytes: Completion/Termination (N= 107, 14) | 0.010 [-0.050 to 0.080] | 0.060 [-0.040 to 0.080]
  Neutrophils: Week 2 (N= 108, 17) | -0.165 [-0.870 to 0.540] | 0.060 [-0.490 to 0.420]
  Neutrophils: Week 4 (N= 109, 14) | -0.130 [-0.680 to 0.450] | -0.140 [-0.300 to 0.540]
  Neutrophils: Month 3 (N= 103, 16) | -0.070 [-0.860 to 0.490] | -0.425 [-0.725 to 0.625]
  Neutrophils: Completion/Termination (N= 107, 14) | 0.050 [-0.820 to 0.480] | 0.055 [-0.570 to 1.150]
  Platelets: Week 2 (N= 107, 16) | -1.0 [-21.0 to 25.0] | 13.5 [-6.5 to 34.5]
  Platelets: Week 4 (N= 108, 13) | 2.0 [-19.5 to 22.5] | -8.0 [-18.0 to 7.0]
  Platelets: Month 3 (N= 102, 15) | 1.5 [-21.0 to 21.0] | -3.0 [-24.0 to 17.0]
  Platelets: Completion/Termination (N= 105, 13) | 0.0 [-20.0 to 20.0] | -1.0 [-15.0 to 14.0]
  Leukocytes: Week 2 (N= 108, 17) | -0.185 [-0.910 to 0.560] | 0.030 [-0.550 to 1.080]
  Leukocytes: Week 4 (N= 109, 14) | -0.180 [-0.930 to 0.640] | -0.005 [-0.670 to 0.750]
  Leukocytes: Month 3 (N= 103, 16) | -0.040 [-1.070 to 0.620] | 0.220 [-0.760 to 1.085]
  Leukocytes: Completion/Termination (N= 107, 14) | -0.020 [-0.900 to 0.680] | 0.250 [-0.710 to 1.800]

28. Secondary Outcome: Changes in Hematology Laboratory Assessments From Screening - Hematocrit
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: Percentage red blood cells
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 108 | 17
Percentage red blood cells
  Week 2 (N= 107, 17) | -0.010 [-0.030 to 0.010] | 0.000 [-0.020 to 0.000]
  Week 4 (N= 108, 13) | -0.010 [-0.020 to 0.005] | -0.010 [-0.020 to 0.000]
  Month 3 (N= 102, 16) | 0.000 [-0.020 to 0.010] | 0.000 [-0.020 to 0.010]
  Completion/Termination (N= 106, 14) | 0.000 [-0.010 to 0.020] | -0.005 [-0.030 to 0.030]

29. Secondary Outcome: Changes in Hematology Laboratory Assessments From Screening - Hemoglobin
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 109 | 17
g/L
  Week 2 (N= 108, 17) | -1.0 [-5.0 to 4.0] | 3.0 [-1.0 to 6.0]
  Week 4 (N= 109, 14) | -1.0 [-5.0 to 5.0] | 0.0 [-2.0 to 7.0]
  Month 3 (N= 103, 16) | 1.0 [-3.0 to 8.0] | 3.5 [-1.5 to 8.5]
  Completion/Termination (N= 107, 14) | 2.0 [-4.0 to 6.0] | 4.5 [-6.0 to 9.0]

30. Secondary Outcome: Changes in Hematology Laboratory Assessments From Screening - Erythrocytes
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: TI/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 109 | 17
TI/L
  Week 2 (N= 108, 17) | -0.10 [-0.20 to 0.10] | 0.10 [-0.20 to 0.10]
  Week 4 (N= 109, 14) | 0.00 [-0.20 to 0.20] | 0.00 [-0.20 to 0.10]
  Month 3 (N= 103, 16) | 0.00 [-0.10 to 0.20] | 0.00 [-0.10 to 0.20]
  Completion/Termination (N= 107, 14) | 0.00 [-0.10 to 0.20] | 0.00 [-0.20 to 0.20]

31. Secondary Outcome: Changes in Lipid Panel Assessments From Screening - Cholesterol; High Density Lipoprotein (HDL); Low Density Lipoprotein (LDL); Triglycerides; and Very Low Density Lipoprotein (VLDL)
Time Frame: Screening, week 2, week 4, month 3, study completion/termination
Population: Safety Analysis Set - Subset of participants with both screening visit data and follow on time point data.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Prophylaxis | On-demand
Number analyzed (Participants) | 115 | 17
mmol/L
  Cholesterol: Week 2 (N= 115, 17) | -0.130 [-0.390 to 0.200] | -0.100 [-0.770 to 0.260]
  Cholesterol: Week 4 (N= 114, 14) | -0.050 [-0.470 to 0.240] | -0.190 [-0.780 to 0.120]
  Cholesterol: Month 3 (N= 109, 17) | -0.070 [-0.330 to 0.360] | 0.040 [-0.220 to 0.400]
  Cholesterol: Completion/Termination (N= 114, 15) | -0.015 [-0.340 to 0.320] | 0.080 [-0.400 to 0.480]
  HDL: Week 2 (N= 115, 17) | 0.000 [-0.100 to 0.080] | -0.130 [-0.190 to -0.020]
  HDL: Week 4 (N= 114, 14) | -0.015 [-0.120 to 0.100] | -0.095 [-0.130 to 0.030]
  HDL: Month 3 (N= 109, 17) | 0.010 [-0.110 to 0.100] | -0.020 [-0.130 to 0.050]
  HDL: Completion/Termination (N= 114, 15) | -0.020 [-0.150 to 0.070] | 0.030 [-0.120 to 0.110]
  LDL: Week 2 (N= 114, 17) | -0.070 [-0.330 to 0.170] | -0.090 [-0.650 to 0.000]
  LDL: Week 4 (N= 112, 13) | -0.080 [-0.350 to 0.245] | -0.320 [-0.470 to -0.210]
  LDL: Month 3 (N= 108, 17) | -0.030 [-0.255 to 0.380] | 0.000 [-0.410 to 0.200]
  LDL: Completion/Termination (N= 113, 15) | 0.050 [-0.310 to 0.310] | -0.050 [-0.450 to 0.380]
  Triglycerides: Week 2 (N= 115, 17) | -0.0600 [-0.4200 to 0.2600] | 0.1700 [-0.0100 to 0.3500]
  Triglycerides: Week 4 (N= 114, 14) | -0.0800 [-0.4000 to 0.2300] | 0.1500 [-0.2500 to 0.6200]
  Triglycerides: Month 3 (N= 109, 17) | -0.1600 [-0.4700 to 0.2100] | 0.3600 [0.2000 to 0.5200]
  Triglycerides: Completion/Termination (N= 114, 15) | 0.0000 [-0.3800 to 0.2300] | 0.1200 [-0.0400 to 0.2100]
  VLDL: Week 2 (N= 114, 17) | -0.0150 [-0.1900 to 0.1200] | 0.0800 [0.0000 to 0.1600]
  VLDL: Week 4 (N= 112, 13) | -0.0350 [-0.1800 to 0.1050] | 0.0400 [-0.1100 to 0.2400]
  VLDL: Month 3 (N= 108, 17) | -0.0700 [-0.2250 to 0.0950] | 0.1600 [0.0900 to 0.2400]
  VLDL: Completion/Termination (N= 113, 15) | 0.0000 [-0.1700 to 0.1000] | 0.0600 [-0.0200 to 0.1000]

ADVERSE EVENTS:
Time Frame: From first exposure to BAX 855 until the end of the study, [at least 50 exposure days or 6 months (±2 weeks), whichever occurs last, for the prophylaxis arm; and 6 months (± 2 weeks) for the on-demand arm].
Description: All study participants were analyzed in a single arm/group.
Groups:
- All Study Participants: All study participants were analyzed in a single arm/group.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 5/137
Other Adverse Events (participants affected / at risk) | 26/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=137)
HERPES ZOSTER INFECTION NEUROLOGICAL (Infections and infestations) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=137)
Nasopharyngitis (Infections and infestations) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 9 (10)
Headache (Nervous system disorders) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per individual PI, but contain common elements. For this study, PIs may be restricted from independently publishing results without prior approval.